CLINICAL TRIAL: NCT06674148
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Study of the Efficacy and Safety of Qifangfeixian Granules in the Treatment of Connective Tissue Disease-Associated Interstitial Lung Disease (CTD-ILD)
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Huilan Zhang (Other)
Responsible Party: Sponsor-Investigator, Huilan Zhang, Professor of department of respiratory and critical care medicine, tongji hospital, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Zhang huilan
Record Dates: First submitted 2024-10-28; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-10

CONDITIONS: Interstitial Lung Disease; Qifangfeixian Granules
Keywords: interstitial lung disease; Qifangfeixian granules
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Intervention Model Description: This is a randomized, placebo-controlled, multicenter study to evaluate the efficacy and safety of Qifangfeixian granules in the treatment of patients with fibrotic interstitial lung disease. The study drugs included Qi fangfeixian Granule and placebo, which was identical in appearance, taste and weight with Qifangfeixian Granule, and were given 1 bag twice a day. This study planned to enroll 124 subjects, who were randomly assigned at a ratio of 1:1, with 62 subjects in each group. Subjects who met all the inclusion criteria at baseline and did not meet the exclusion criteria were randomized to either of the following two groups: (1) Qifangfeixian Granule treatment group: oral administration of Qifangfeixian granule, 1 bag, 2 times a day; (2) Placebo (PRO) control group: oral administration of placebo, 1 bag, 2 times a day. Patients were evaluated after 12 weeks of treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Qifangfeixian granule group (Experimental): 62 cases in the group , 2 times a day, each time 1 bag of Qifangfeixian granules, oral administration
  Interventions: Drug: Qifangfeixian granules
- Placebo control group (Placebo Comparator): 62 control group patients were orally administered with 1 bag of placebo twice a day
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Qifangfeixian granules — The experimental group was treated with Qifangfixian granules
  Arms: Qifangfeixian granule group
Other: Placebo — The control group was treated with placebo
  Arms: Placebo control group

SUMMARY:
Interstitial lung disease (ILD) is a heterogeneous group of diseases characterized by inflammation and/or fibrinization of the alveolar unit due to a variety of known or unknown causes. CTD-ILD is one of its common categories and includes any ILD with a definite diagnosis of connective tissue disease or with a set of symptoms, signs, and abnormalities suggested by laboratory examination. The incidence of CTD-ILD varies from home to abroad. Foreign studies indicate that the number of CTD-ILD in this study accounted for 34.8% of the total number of ILD in this study, while domestic studies indicate that the number of CTD-ILD in this study accounted for 67% of the total number of ILD. At present, the treatment of CTD-ILD includes hormone, immunosuppressant cyclophosphamide, mortemycophenate, tacrolimus, etc. The above treatment has great side effects, which may increase the risk of infection and the incidence of malignant tumor. Traditional Chinese medicine has unique advantages in alleviating the clinical symptoms of the disease, reducing the use of hormones and hormone complications, and preventing infection. Qifangfeixian granule is derived from "Fangji Huangqi Decoction" in the Summary of Golden Chamber. Modern pharmacology shows that Huangqi has the functions of regulating immunity, protecting liver, antibacterial and antiviral, etc. In order to further evaluate the effectiveness and safety of using Qifangfeixian granule (Huangqi, Fangji, dogwood, dodder, ginkgo, salvia miltiorrhizae, Taoren, etc.) in the treatment of CTD-ILD patients, Determined to explore a path of CTD-ILD treatment with Chinese characteristics, we hereby apply for a multicenter controlled clinical study.

DETAILED DESCRIPTION:
ILD is a common complication of CTD, with high disability rate and fatality rate, poor prognosis and high fatality rate. Ild is one of the main causes threatening the life of patients. The objective of this study was to evaluate the efficacy and safety of Qifangfeixian granules in the treatment of CTD-ILD patients, and to provide a new treatment plan for CTD-ILD patients. This is a randomized, placebo-controlled, multicenter study to evaluate the efficacy and safety of Qifangfeixian granules in the treatment of patients with fibrotic interstitial lung disease. The study drugs included Qifangfeixian Granule and placebo, which was identical in appearance, taste and weight with Qifangfeixian Granule, and were given 1 bag twice a day. This study planned to enroll 124 subjects, who were randomly assigned at a ratio of 1:1, with 62 subjects in each group. Subjects who met all the inclusion criteria and did not meet the exclusion criteria at baseline were randomly assigned to either of the following two groups: (1) Qifangfeixian Granule treatment group: orally administered with 1 bag of Qifangfeixian granule twice a day; (2) Placebo (PRO) control group: orally administered with 1 bag of placebo twice a day. If participants withdraw from the study early, they will be followed up for 4 weeks. Participants were allowed to make dose adjustments during treatment and were withdrawn from the study when a serious adverse event occurred or medication was discontinued due to an adverse event. Throughout the course of the study, safety checks and assessments will be conducted according to the time points specified in the protocol, including adverse events, HRCT, clinical laboratory tests (blood routine, blood biochemistry, urine routine, coagulation function, myocardial enzymes, etc.), 12-lead electrocardiogram, vital signs, and physical examination. Patient data were recorded on the case report form based on the visit.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or female aged 18-80. 2. Both conditions (1) and (2) are met or conditions (3) are met:

  1. Diagnosis of CTD: CTD can be clearly diagnosed by referring to the classification criteria of each disease. SLE, SS, SSc, RA, PM/DM, etc. can be diagnosed according to the corresponding international classification standards.
  2. Diagnosis of ILD: Combined with the patient's symptoms such as progressive dyspnea, dry cough, pulmonary signs such as Velcro rales in both lungs, pulmonary function examination suggesting restrictive ventilation disorder and diffusion dysfunction, High-resolution CT of the chest indicated diffuse nodules, ground-glass changes, alveolar consolidation, thickening of interlobular septum, downline pleura, mesh shadows with cyst formation or cellular changes, tractive bronchiectasis, or structural changes of the lung.
  3. ILD (confirmed by high-resolution chest CT or surgical lung biopsy) is present, and ① other known etiology is excluded; ② A definite CTD cannot be diagnosed; (3) At least 2 of the following 3 characteristics: A. Clinical manifestations: (1) distal finger skin cracks (" technician hand "); (2) distal fingertip skin ulcer; (3) Inflammatory arthritis or polyjoint stiffness ≥60 min; (4) telangiectasia of the palm or finger abdomen; (5) Reynolds phenomenon; (6) unexplained swelling of the fingers; (7) Unexplained fixed rash of extended fingers (Gottron sign).

B. Serological manifestations: (1) ANA titer ≥ 1:320, diffuse type, spot type, homogeneous type, or ①ANA nucleolar type (arbitrary titer), or ②ANA centromere type (arbitrary titer); (2) Rheumatoid factor ≥2 times the upper limit of normal reference value; (3) Positive anti-CCP antibody; (4) Anti-double-stranded DNA antibody is positive; (5) Anti-SSA (Ro) antibody positive; (6) Anti-SSB (La) antibody positive; (7) Positive anti-ribonucleoprotein antibody; (8) Positive anti-SM antibody; (9) Anti-topoisomerase (Scl-70) antibody was positive; (10) Anti-TRNA synthase (such as Jo-l, PL-7, PL-12; Others include EJ, 0J, KS, Zo, tRS) antibody positive; (11) Anti-PM-SCL antibody is positive; (12) Anti-melanoma differentiation related gene 5 (MDA5) antibody was positive.

C. Morphological findings: (1) Chest high-resolution CT findings: ①NSIP, or ②OP, or ③NSIP overlapping OP, or ④LIP; (2) Pathological types of surgical lung biopsy: ①NSIP, or ②OP, or ③NSIP overlapping OP, or ④LIP, or ⑤ interstitial lymphocyte infiltration associated with hair center formation, or ⑥ diffuse lymphoplasmic cell infiltration (with or without lymphofollicular formation); (3) Multiple thoracic involvement (except interstitial pneumonia) : ① unexplained pleural effusion/pleural thickening; ② Unexplained pericardial effusion/pericardial thickening; (3) Endogenous airway diseases of unknown origin, including airflow obstruction, bronchiolitis, or bronchiectasis (confirmed by pulmonary function, imaging, or histopathology); ④ Pulmonary vascular disease of unknown cause.

Exclusion Criteria:

* 1. When visiting 1, set AST and ALT to 1.5x ULN 2. Bilirubin > 1.5 x ULN at visit 1 3. At visit 1, creatinine clearance was < 30 mL/min as calculated by Cockcroft - Gault formula.

  4. Patients with underlying chronic liver disease (Child Pugh A, B, or C liver injury).

  5. Received other investigational medications within 1 month or 6 half-lives (whichever is greater) prior to the screening visit (visit 1).

  6. Significant pulmonary arterial hypertension (PAH) as defined by any of the following criteria: (1) clinical/echocardiographic evidence of prior significant right heart failure; (2) Medical history, including the right cardiac catheter showing cardiac index ≤2L/min/m2; (3) parenteral administration of eprostol/traprostacycline is required to treat PAH.

  7. Other lung abnormalities deemed clinically significant by the investigators. 8. Major extrapulmonary physical limitations (e.g., chest wall malformations, massive pleural effusion).

  9. Cardiovascular disease, any of the following: (1) severe hypertension within 6 months of visit 1, uncontrollable after treatment (≥160/100 mmHg); (2) myocardial infarction within 6 months of visit 1; (3) Unstable angina pectoris within 6 months of visit 1 10. History of severe central nervous system (CNS) events. 11. Known allergy to the experimental drug. 12. Other medical conditions that may interfere with the testing procedure or, as determined by the investigator, may interfere with trial participation or may put the patient at risk when participating in the trial.

  13. Women in this trial who are pregnant, breastfeeding or planning to become pregnant.

  14. Patients were unable to understand or follow trial procedures, including completing questionnaires on their own without assistance.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2024-10-25 (Actual); Primary Completion 2027-05-20 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
forced vital capacity(FVC) | 12 weeks
  Changes of FVC (ml) from baseline in the experimental group and the control group after 12 weeks of treatment with Qifangfeixian granules

SECONDARY OUTCOMES:
hormone dosage change | 12 weeks
  Changes of hormone dosage from baseline in the experimental group and the control group after 12 weeks of treatment with Qifangfeixian granules
Pulmonary fibrosis survival symptom score | 12 weeks
  Change of pulmonary fibrosis survival symptom score from baseline after 12 weeks of treatment with Qifangfeixian granules in experimental group and control group using L-PF questionnaire.

OTHER OUTCOMES:
dyspnea scores | 12 weeks
  Percentage decrease in dyspnea score from baseline after 12 weeks of treatment with Qifangfeixian granules in experimental group compared with control group
Forced expiratory volume in one second(FEV1) | 12 weeks
  Percentage decrease in FEV1 from baseline after 12 weeks of treatment with Qifangfeixian granules in the experimental group compared with the control group
Chest CT | 12 weeks
  Percentage decrease in chest CT score from baseline after 12 weeks of treatment with Qifangfeixian granules in experimental group compared with control group
Combined infection and acute exacerbation | 12 weeks
  Evaluation of infection and acute exacerbation after 12 weeks of treatment with Qifangfeixian granules in experimental group and control group
Hospitalization or death from respiratory causes | 12 weeks
  Time between trial and hospitalization or death due to respiratory causes in the experimental group compared with the control group

CONTACTS AND LOCATIONS:
Overall Officials: Zhang Huilan, PD, Study Chair — Tongji hospital affiliated to huazhong university of science and technology, Wuhan, hubei
Locations (1):
- Tongji hospital affiliated to huazhong university of science and technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] An L, Peng LY, Sun NY, Yang YL, Zhang XW, Li B, Liu BL, Li P, Chen J. Tanshinone IIA Activates Nuclear Factor-Erythroid 2-Related Factor 2 to Restrain Pulmonary Fibrosis via Regulation of Redox Homeostasis and Glutaminolysis. Antioxid Redox Signal. 2019 May 20;30(15):1831-1848. doi: 10.1089/ars.2018.7569. Epub 2018 Sep 22. PMID 30105924
- [Background] Yang CG, Mao XL, Wu JF, An X, Cao JJ, Zhang XY, Li M, Zhang FF. Amelioration of Lung Fibrosis by Total Flavonoids of Astragalus via Inflammatory Modulation and Epithelium Regeneration. Am J Chin Med. 2023;51(2):373-389. doi: 10.1142/S0192415X23500192. Epub 2023 Jan 20. PMID 36655684
- [Background] You Zaijing, Synopsis of Golden Chamber (in Chinese). Beijing: China Traditional Chinese Medicine Press, 2006:11
- [Background] Wilson TM, Solomon JJ, Demoruelle MK. Treatment approach to connective tissue disease-associated interstitial lung disease. Curr Opin Pharmacol. 2022 Aug;65:102245. doi: 10.1016/j.coph.2022.102245. Epub 2022 Jun 1. PMID 35662004
- [Background] Li L, Zuo X, Luo H, Li Y, You Y, Duan L, Zhang W, Zhao H, Li T, Ning W, Xie Y, Liu S, Xie X, Jiang Y, Wu S, Zhu H, Zhou Y. Mortality trend of inpatients with connective tissue diseases: 2005-2014. Zhong Nan Da Xue Xue Bao Yi Xue Ban. 2017 Aug 28;42(8):927-933. doi: 10.11817/j.issn.1672-7347.2017.08.009. PMID 28872084
- [Background] Spagnolo P, Distler O, Ryerson CJ, Tzouvelekis A, Lee JS, Bonella F, Bouros D, Hoffmann-Vold AM, Crestani B, Matteson EL. Mechanisms of progressive fibrosis in connective tissue disease (CTD)-associated interstitial lung diseases (ILDs). Ann Rheum Dis. 2021 Feb;80(2):143-150. doi: 10.1136/annrheumdis-2020-217230. Epub 2020 Oct 9. PMID 33037004
- [Background] Yang Xiguang, Chen Weisong, Xu Jilin, et al. Analysis of clinical features of interstitial lung disease associated with connective tissue disease in 186 cases. Chinese Journal of General Practitioners, 2019,18 (3) : 250-250.
- [Background] Zou Qing-Hua, Lu Yue-Wu, ZHOU Jing-Guo, et al. Diagnosis and treatment of interstitial lung disease associated with connective tissue disease. Chinese Journal of Internal Medicine, 2002, 61(11) : 1217-1223.
- [Background] Alhamad EH. Interstitial lung diseases in Saudi Arabia: A single-center study. Ann Thorac Med. 2013 Jan;8(1):33-7. doi: 10.4103/1817-1737.105717. PMID 23440334
- [Background] Aithala R, Alex AG, Danda D. Pulmonary hypertension in connective tissue diseases: an update. Int J Rheum Dis. 2017 Jan;20(1):5-24. doi: 10.1111/1756-185X.13001. Epub 2017 Feb 16. PMID 28205373
- [Background] Mathai SC, Danoff SK. Management of interstitial lung disease associated with connective tissue disease. BMJ. 2016 Feb 24;352:h6819. doi: 10.1136/bmj.h6819. PMID 26912511
- [Background] Wijsenbeek M, Cottin V. Spectrum of Fibrotic Lung Diseases. N Engl J Med. 2020 Sep 3;383(10):958-968. doi: 10.1056/NEJMra2005230. No abstract available. PMID 32877584
- [Background] Wijsenbeek M, Suzuki A, Maher TM. Interstitial lung diseases. Lancet. 2022 Sep 3;400(10354):769-786. doi: 10.1016/S0140-6736(22)01052-2. Epub 2022 Aug 11. PMID 35964592